CLINICAL TRIAL: NCT04052789
Title: Clinical Evaluation of Internal Fit of Milled BioHPP Polyetheretherketone (PEEK) - Based Versus Zirconia-Based Single Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Gamal Adly, Resident, Fixed Prosthodontices Department,Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-08-03
Record Dates: First submitted 2019-08-04; First posted 2019-08-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Badly Decayed Teeth andTeeth Restored With Large Filling Restorations and Endodontically Treated Teeth and Malformed Teeth and Malposed Teeth
MeSH Terms: conditions — Tooth, Nonvital; Tooth Abnormalities | interventions — Composite Resins

STUDY DESIGN:
Masking Description: Double(participant, outcome Assessor) Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia single posterior crowns veneered with ceramics (Active Comparator): 'In the first visit, a Face-to-Face adherence session will be held in which the patient should be informed about the study steps and how to maintain oral hygiene measures. Further sessions will occur at the follow-up visits
  Interventions: Other: BioHPP PEEK copings veneered with composite resin
- BioHpp PEEK single posterior crowns veneered with compos (Experimental): In the first visit, a Face-to-Face adherence session will be held in which the patient should be informed about the study steps and how to maintain oral hygiene measures. Further sessions will occur at the follow-up visits
  Interventions: Other: BioHPP PEEK copings veneered with composite resin

INTERVENTIONS:
Other: BioHPP PEEK copings veneered with composite resin — In the first visit, a Face-to-Face adherence session will be held in which the patient should be informed about the study steps and how to maintain oral hygiene measures. Further sessions will occur at the follow-up visits . Participant patients will be asked about any problems they are having. Patients will be recalled every two months for one year for follow up visits.

SUMMARY:
All ceramic crowns are indicated in case of mild to moderate discoloration, restoration of traumatized or fractured teeth and abnormal tooth anatomy. The success of dental restorations is determined by four main factors: biocompatibility, aesthetic value, resistance to fracture and marginal adaptation. . An inadequate marginal fit may compromise the longevity of the restoration since cement film exposure to the oral environment can lead to its dissolution . .

Polyetheretherketone (PEEK) is a polymer that has many potentials uses in dentistry. Polyetheretherketone (PEEK) can be used to support fixed dental prostheses. However, information about physio mechanical characterization is still scarce.

Aim of the study:

- The aim of this study is to evaluate the internal fit of milled BioHPP PEEK-based versus zirconia-based single crowns.

ELIGIBILITY:
Inclusion Criteria:

* From 18-50 years old, be able to read and sign the informed consent document.
* Patient Have no active periodontal or pulpal diseases, have teeth with good restorations
* Patient Psychologically and physically able to withstand conventional dental procedures
* Patients with teeth problems indicated for single posterior crowns:

Exclusion Criteria:

* Patient less than 18 or more than 50 years
* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene and uncooperative patients
* Patients in the growth stage with partially erupted teeth
* Patient with Psychiatric problems or unrealistic expectations
* Patient with Lack of opposing dentition in the area of interest

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Internal fit of the crown by measuring the thickness of the replica by steriomicroscope | one year
  measured by replica technique and steriomicroscope

SECONDARY OUTCOMES:
secondary caries if present at the margin of the crown by using probe | one year
  Measured by modified Ryge criteria Alpha (A)The restoration is a continuation of existing anatomic form adjacent to the restoration.
  Bravo (B)There is visual evidence of dark keep discoloration adjacent to the restoration (but notAlpha (A)The restoration is a continuation of existing anatomic form adjacent to the restoration.
  Bravo (B)There is visual evidence of dark keep discoloration adjacent to the restoration (but not directly associated with cavosurface margins).
  directly associated with cavosurface margins).

OTHER OUTCOMES:
patient satisfaction | one year
  Measured by VAS(questionnaire)Numerical (discrete) ("0" unsatisfied - "10" satisfied)

IPD SHARING:
Plan to Share IPD: Undecided